CLINICAL TRIAL: NCT04319900
Title: Clinical Trial of Favipiravir Tablets Combine With Chloroquine Phosphate in the Treatment of Novel Coronavirus Pneumonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Lihong Liu, Prof., Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-K-24-2
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Novel Coronavirus Pnuemonia
MeSH Terms: interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- favipiravir tablets+chloroquine phosphatetablets tablets group (Experimental): favipiravir tablets+chloroquine phosphatetablets tablets
  Interventions: Drug: favipiravir tablets+chloroquine phosphatetablets tablets
- favipiravir tablets group (Experimental): favipiravir tablets
  Interventions: Drug: Favipiravir tablets
- placebo treatment group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: favipiravir tablets+chloroquine phosphatetablets tablets — Favipiravir tablets+ chloroquine phosphate tablets group: 50 patients (anticipated).
  Favipiravir tablets: On the first day, once for 1600 mg, twice a day; From the 2nd day to the 10th day, once for 600 mg, twice a day; maximum of 10 days for oral administration of the drug.
  Chloroquine phosphate tablets: a total of 1000mg split into two times on day one; from day two to day three, 500mg, once a day; from day four to day ten, 250mg, once a day. Maximum of 10 days for oral administration of the drug.
  Arms: favipiravir tablets+chloroquine phosphatetablets tablets group
Drug: Favipiravir tablets — Favipiravir tablets group: 50 patients (anticipated). Favipiravir tablets: On the first day, once for 1600 mg, twice a day; From the 2nd day to the 10th day, once for 600 mg, twice a day; maximum of 10 days for oral administration of the drug.
  Arms: favipiravir tablets group
Drug: Placebo — Placebo for favipiravir tablets is produced by Zhejiang Haizheng pharmaceutical co, LTD, batch no. 21812252, Placebo for chloroquine phosphate tablets is produced by the Chinese people's liberation army academy of military science military medical research institute production, batch no. 20200215. All placebos were complied with the quality inspection standard.
  Arms: placebo treatment group

SUMMARY:
This study is a multi-centered, three-armed, randomized, double-blinded, controlled study, namely, the oral trial drug favipiravir tablets plus chloroquine phosphatetablets tablets group (combined group), the oral trial drug favipiravir tablets group (pirovir group), and the oral placebo treatment group (control group). The total number of enrolled cases in this study was set at 150.

During the treatment, the clinical data of the subjects were collected, the changes of viral load and biochemical indicators were detected, and the outcome of the subjects was monitored.

The main indicators of efficacy include improvement or recovery of respiratory symptoms and viral nucleic acid shedding. The rate of progression to severe disease, duration of fever, peripheral blood index and improvement time of pulmonary imaging were the secondary indicators to evaluate the efficacy.

Statistical analysis was performed at the middle and final stages of the study to evaluate the efficacy and safety of favipiravir tablets combined with chloroquine phosphatetablets tablets in the treatment of novel coronavirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18-75 years old
* Patients previously diagnosed with novel coronavirus pneumonia: the course of illness is no more than 14 days; if the course of the disease was more than 14 days, patient meets one of the following conditions can also be included in the group: (1) No apparent absorption or progression of chest radiograph was observed within 7 days; (2) respiratory symptoms (chest tightness, or cough, or breathing difficulties); (3) Test for viral nucleic acid positive within 3 days.
* informed consent should be signed by the participate or an authorized agent
* Agree to clinical samples collection
* Female or male subjects of childbearing age agree to take effective contraceptive measures within 3 months of the last oral medication to ensure that female or male partners of childbearing age do not become pregnant

Exclusion Criteria:

* Severe vomiting or difficulty ingesting medication
* Woman who are pregnant or during lactation
* Patients received lopinavir/ridonavir, ribavirin, interferon and monoclonal antibody specific antiviral drugs three days before enrollment
* Cases of respiratory failure requiring mechanical ventilation
* Shock
* Combined with other organ failure and requires ICU care
* Clinical prognostic non-survival, palliative care, or in deep coma and no have response to supportive treatment within three hours of admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-25 (Estimated)

PRIMARY OUTCOMES:
Time of Improvement or recovery of respiratory symptoms | 10 days during the intervention period
  Time of improvement or recovery of respiratory symptoms
Number of days virus nucleic acid shedding | 10 days during the intervention period
  Number of days from positive to negative for test of swab or sputum virus nucleic acid
Frequency of Improvement or recovery of respiratory symptoms | 10 days during the intervention period
  Frequency of improvement or recovery of respiratory symptoms

SECONDARY OUTCOMES:
Duration of fever | 10 days during the intervention period
  Duration of fever after recruitment
Frequencies of progression to severe illness | 10 days during the intervention period
  Disease is defined as severe if it meets any of the following criteria: 1.Respiratory rate ≥30/min; 2. Oxygen saturation ≤93%; 3. Arterial partial oxygen pressure (PaO2)/oxygen absorption concentration (FiO2) ≤300 mmHg (1 mmHg=0.133 kPa)
Time of improvement of pulmonary imaging | 10 days during the intervention period
  Time of improvement of pulmonary imaging
Peripheral blood c-reactive protein concentration | day-1,3,7,14 after the intervention period
  Peripheral blood c-reactive protein concentration
Absolute value of peripheral blood lymphocytes | day-1,3,7,14 after the intervention period
  Absolute value of peripheral blood lymphocytes
percentage of peripheral blood lymphocytes | day-1,3,7,14 after the intervention period
  percentage of peripheral blood lymphocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang hospital, Beijing, Beijing Municipality, China